CLINICAL TRIAL: NCT05342129
Title: Effects of Exercise Intervention on Muscle Strength in Severely Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020-07-022B
Record Dates: First submitted 2022-03-02; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Intensive Care Unit Patients
Keywords: Intensive care unit patients, exercise Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise bike (Experimental): exercise is to use an exercise bike, start pedaling on the first day, time setting: 20 minutes, speed: 2, and adopt passive mode. If you can complete the exercise on the first day, the time will be adjusted to 30 minutes on the second day. If you cannot complete the exercise on the first day, the time will still start from 20 minutes on the second day. The maximum time is 30 minutes. If you can complete 30 minutes of passive exercise for 3 consecutive days, the fourth day will be adjusted to active exercise. The entire exercise training is seven days a week, once a day, once a 30-minute, at least 5 days. Those who were discharged to the general ward continued to complete this exercise training for up to 28 days.
  Interventions: Other: exercise bike
- regular rehabilitation exercises (No Intervention): walking exercise

INTERVENTIONS:
Other: exercise bike — exercise is to use an exercise bike, start pedaling on the first day, time setting: 20 minutes, speed: 2, and adopt passive mode. If you can complete the exercise on the first day, the time will be adjusted to 30 minutes on the second day. If you cannot complete the exercise on the first day, the time will still start from 20 minutes on the second day. The maximum time is 30 minutes. If you can complete 30 minutes of passive exercise for 3 consecutive days, the fourth day will be adjusted to active exercise. The entire exercise training is seven days a week, once a day, once a 30-minute, at least 5 days. Those who were discharged to the general ward continued to complete this exercise training for up to 28 days.
  Arms: exercise bike

SUMMARY:
In recent years, due to the improvement in the survival rate of the intensive care unit, the problem of severe systemic fatigue (Intensive care unit acquired weakness; ICUAW) has continued to receive attention. Muscle mass decreases by 3-11% within a week, resulting in decreased muscle strength and muscle atrophy. Current studies suggest that ICUAW can lead to poorer function, prolonged ICU stay, and decreased quality of life.

This study aimed to understand the muscle strength of critically ill patients and to explore the effect of exercise intervention on improving muscle strength. The experimental group received a four-week exercise bike intervention plus conventional rehabilitation exercises, while the control group received conventional rehabilitation exercises.

DETAILED DESCRIPTION:
The content of the exercise is to use an exercise bike, start pedaling on the first day, time setting: 20 minutes, speed: 2, and adopt passive mode. If you can complete the exercise on the first day, the time will be adjusted to 30 minutes on the second day. If you cannot complete the exercise on the first day, the time will still start from 20 minutes on the second day. The maximum time is 30 minutes. If you can complete 30 minutes of passive exercise for 3 consecutive days, the fourth day will be adjusted to active exercise. The entire exercise training is seven days a week, once a day, once a 30-minute, at least 5 days. Those who were discharged to the general ward continued to complete this exercise training for up to 28 days. Stop exercising if heartbeat > 140, mean arterial pressure < 65, blood oxygen < 90%, respiration > 35 beats/min, or the patient requests to stop during exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 20 years old
2. Conscious
3. willing to participate in this study, and signed the consent form
4. no lower extremity activity taboo, and can walk independently before admission

Exclusion Criteria:

1. Have neuromuscular disease.
2. Unable to step on a bed bike.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Basic Demographic Health Assessment Form | baseline
  Age, sex, diagnosis, disease severity, reason for ICU admission
days in intensive care unit | baseline
  Health Assessment Form
days on ventilator | baseline
  Health Assessment Form
total days in hospital | baseline
  Health Assessment Form
body mass index | baseline
  Health Assessment Form
level of albumin | baseline
  Health Assessment Form
The daily observation record sheet includes | up to 28 days
  Vital signs,respirator is used or not,bicycle use pattern,speed and time,reasons for stopping

SECONDARY OUTCOMES:
Hand grip strength | baseline(T0)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 3 days after intervention(T1)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 7 days after intervention(T2)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 10 days after intervention(T3)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 14 days after intervention(T4)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 17 days after intervention(T5)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 21 days after intervention(T6)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
Hand grip strength | 28 days after intervention(T7)
  Using a Grip Strength Tester to Measure Dominant Hand Muscle Strength
foot lift | baseline(T0)
  Use a tape to measure foot lift
foot lift | 3 days after intervention(T1)
  Use a tape to measure foot lift
foot lift | 7days after intervention(T2)
  Use a tape to measure foot lift
foot lift | 10days after intervention(T3)
  Use a tape to measure foot lift
foot lift | 14days after intervention(T4)
  Use a tape to measure foot lift
foot lift | 17ays after intervention(T5)
  Use a tape to measure foot lift
foot lift | 21days after intervention(T6)
  Use a tape to measure foot lift
foot lift | 28days after intervention(T7)
  Use a tape to measure foot lift
walking distance in 6 minutes | baseline(T0)
  Measure 6-minute walking distance
walking distance in 6 minutes | 3 days after intervention(T1)
  Measure 6-minute walking distance
walking distance in 6 minutes | 7 days after intervention(T2)
  Measure 6-minute walking distance
walking distance in 6 minutes | 10days after intervention(T3)
  Measure 6-minute walking distance
walking distance in 6 minutes | 14days after intervention(T4)
  Measure 6-minute walking distance
walking distance in 6 minutes | 17days after intervention(T5)
  Measure 6-minute walking distance
walking distance in 6 minutes | 21days after intervention(T6)
  Measure 6-minute walking distance
walking distance in 6 minutes | 28ays after intervention(T7)
  Measure 6-minute walking distance

CONTACTS AND LOCATIONS:
Overall Officials: Tao-Fen Hsiung, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- TaipeiVGH, Taipei, Taipei City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Result] Camargo Pires-Neto R, Fogaca Kawaguchi YM, Sayuri Hirota A, Fu C, Tanaka C, Caruso P, Park M, Ribeiro Carvalho CR. Very early passive cycling exercise in mechanically ventilated critically ill patients: physiological and safety aspects--a case series. PLoS One. 2013 Sep 9;8(9):e74182. doi: 10.1371/journal.pone.0074182. eCollection 2013. PMID 24040200
- [Result] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Result] Eggmann S, Verra ML, Luder G, Takala J, Jakob SM. Effects of early, combined endurance and resistance training in mechanically ventilated, critically ill patients: A randomised controlled trial. PLoS One. 2018 Nov 14;13(11):e0207428. doi: 10.1371/journal.pone.0207428. eCollection 2018. PMID 30427933
- [Result] Hermans G, Van Mechelen H, Clerckx B, Vanhullebusch T, Mesotten D, Wilmer A, Casaer MP, Meersseman P, Debaveye Y, Van Cromphaut S, Wouters PJ, Gosselink R, Van den Berghe G. Acute outcomes and 1-year mortality of intensive care unit-acquired weakness. A cohort study and propensity-matched analysis. Am J Respir Crit Care Med. 2014 Aug 15;190(4):410-20. doi: 10.1164/rccm.201312-2257OC. PMID 24825371
- [Result] Kho ME, Molloy AJ, Clarke FJ, Ajami D, McCaughan M, Obrovac K, Murphy C, Camposilvan L, Herridge MS, Koo KK, Rudkowski J, Seely AJ, Zanni JM, Mourtzakis M, Piraino T, Cook DJ; Canadian Critical Care Trials Group. TryCYCLE: A Prospective Study of the Safety and Feasibility of Early In-Bed Cycling in Mechanically Ventilated Patients. PLoS One. 2016 Dec 28;11(12):e0167561. doi: 10.1371/journal.pone.0167561. eCollection 2016. PMID 28030555
- [Result] Kho ME, Molloy AJ, Clarke FJ, Reid JC, Herridge MS, Karachi T, Rochwerg B, Fox-Robichaud AE, Seely AJ, Mathur S, Lo V, Burns KE, Ball IM, Pellizzari JR, Tarride JE, Rudkowski JC, Koo K, Heels-Ansdell D, Cook DJ. Multicentre pilot randomised clinical trial of early in-bed cycle ergometry with ventilated patients. BMJ Open Respir Res. 2019 Feb 18;6(1):e000383. doi: 10.1136/bmjresp-2018-000383. eCollection 2019. PMID 30956804
- [Result] Machado ADS, Pires-Neto RC, Carvalho MTX, Soares JC, Cardoso DM, Albuquerque IM. Effects that passive cycling exercise have on muscle strength, duration of mechanical ventilation, and length of hospital stay in critically ill patients: a randomized clinical trial. J Bras Pneumol. 2017 Mar-Apr;43(2):134-139. doi: 10.1590/S1806-37562016000000170. PMID 28538781